CLINICAL TRIAL: NCT02336763
Title: Prophylactic Hepatic Irradiation for Uveal Melanoma
Brief Title: Radiation Therapy in Preventing Liver Metastases in Patients With Uveal Melanoma Who HaveMonosomy 3 or DecisionDx Class 2 Disease and Are More Likely to Develop Liver Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed due to lack of accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-000903; NCI-2014-02254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID466 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2016-03

CONDITIONS: Iris Melanoma; Medium/Large Size Posterior Uveal Melanoma; Stage IIA Uveal Melanoma; Stage IIB Uveal Melanoma; Stage IIIA Uveal Melanoma; Stage IIIB Uveal Melanoma; Stage IIIC Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (external beam radiation therapy) (Experimental): Patients undergo external beam radiation therapy daily over 20 minutes on Monday-Friday for up to 10 fractions over approximately 2 weeks.
  Interventions: Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam RT
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies giving radiation therapy to the liver in patients with uveal (eye) melanoma who have a specific chromosome loss (monosomy 3) or are DecisionDx Class 2 and therefore more likely to have their disease spread from the eye to the liver. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Early radiation to the liver may reduce the development of tumors in the liver and the overall risk of disease recurrence.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Progression free survival in patients treated with prophylactic hepatic irradiation.

SECONDARY OBJECTIVES:

I. Acute and late term toxicity and overall survival.

OUTLINE:

Patients undergo external beam radiation therapy daily over 20 minutes on Monday-Friday for 10 fractions over approximately 2 weeks.

After completion of study treatment, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed uveal melanoma
* Monosomy 3 status (by fluorescent in situ hybridization [FISH] or multiplex ligation-dependent probe amplification [MLPA]) or DecisionDx class 2
* Tumor thickness > 3.0 mm
* Has received definitive treatment of uveal melanoma with brachytherapy, proton therapy, stereotactic radiosurgery, or enucleation
* Karnofsky performance status (KPS) >= 70 or Eastern Cooperative Oncology Group (ECOG)
* Total bilirubin < 1.5 mg/dl
* Aspartate transaminase (AST) up to two times normal limit
* Alanine transaminase (ALT) up to two times normal limit
* Creatinine < 2.0 mg/dl
* Functional left kidney based on computed tomography (CT) imaging
* Positron emission tomography (PET)/CT demonstrating no evidence of metastatic disease
* If a woman is of childbearing potential, a negative serum pregnancy test must be documented; women of childbearing potential must agree to use contraception for the duration of radiation therapy (approximately 3 weeks)
* Understands the trial and procedures and is willing and able to sign the Informed Consent Form

Exclusion Criteria:

* Previous malignancy, other than localized cutaneous squamous cell carcinoma or basal cell carcinoma
* History of prior irradiation to the thorax or abdomen
* Inadequate hepatic or kidney function (as specified above)
* Active peptic ulcer disease
* Upper gastrointestinal bleeding
* Pregnant women or women that refuse to use contraception throughout the entire study period
* Currently receiving chemotherapy
* Refuses to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Kamrava, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (External Beam Radiation Therapy)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: only two subjects were enrolled
Arm/Group | Treatment (External Beam Radiation Therapy)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Time Frame: Up to 5 years
Population: Study terminated early no analysis conducted. Subjects would need to be followed for up to 5 years to answer this objective. Subject 1 was followed 5 months and subject 2 was followed 2 months. Therefore, data was not collected from any subject for this Outcome Measure.
Arm/Group | Treatment (External Beam Radiation Therapy)
Number analyzed (Participants) | 0

2. Primary Outcome: Reduction in Liver Metastasis
Time Frame: Up to 5 years
Population: study terminated early no analysis conducted. Data was not collected from any subject for this Outcome Measure.
Arm/Group | Treatment (External Beam Radiation Therapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Frequency and Severity of Acute Toxicity Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4
Time Frame: Within 3 months of study treatment
Population: study terminated early no analysis conducted. Data was not collected from any subject for this Outcome Measure.
Arm/Group | Treatment (External Beam Radiation Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Frequency and Severity of Late Toxicity Per NCI CTCAE Version 4
Time Frame: More than 3 months after study treatment
Population: study terminated early no analysis conducted. Data was not collected from any subject for this Outcome Measure.
Arm/Group | Treatment (External Beam Radiation Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Time Frame: Up to 5 years
Population: study terminated early no analysis conducted. Data was not collected from any subject for this Outcome Measure.
Arm/Group | Treatment (External Beam Radiation Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Distant Failure Rates
Description: Cumulative incidence approach (Kaplan-Meier [K-M] plots and Cox proportional hazard modeling) will be used to estimate distant failure rates.
Time Frame: Up to 5 years
Population: study terminated early no analysis conducted. Data was not collected from any subject for this Outcome Measure.
Arm/Group | Treatment (External Beam Radiation Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Disease-specific Survival
Description: Cumulative incidence approach (K-M plots and Cox proportional hazard modeling) will be used to estimate disease-specific survival.
Time Frame: Up to 5 years
Population: study terminated early no analysis conducted. Data was not collected from any subject for this Outcome Measure.
Arm/Group | Treatment (External Beam Radiation Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (External Beam Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes